CLINICAL TRIAL: NCT02580942
Title: Efficacy Study of Acupoint Sticking in Treating Winter Diseases in Summer to Treat Asthma of Kidney Yang Deficiency Type
Brief Title: Efficacy Study of Acupoint Sticking in Summer to Treat Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Shanghai Municipal Health Bureau (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13401905400
Record Dates: First submitted 2015-07-30; First posted 2015-10-20 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2015-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupoint sticking therapy group (Experimental): 36 patients receive acupoint sticking treatment of Chinese herbal medicine on Dazhui(GV14) and Tiantu(RN22), and magnetic stickers on Feishu(BL13), Pishu(BL20) and Shenshu(BL23) once every other day, retention for 4 hours. Patients receive verum acupoint sticking therapy once every other day with a total of 18 sessions in 6 weeks.
  Interventions: Device: Magnetic stickers; Drug: Chinese herbal medicine
- Sham sticking therapy group (Sham Comparator): 36 patients receive acupoint sticking treatment of Chinese herbal medicine on Dazhui(GV14) and Tiantu(RN22), and sham magnetic stickers on Feishu(BL13), Pishu(BL20) and Shenshu(BL23) once every other day, retention for 4 hours. Patients receive verum acupoint sticking therapy once every other day with a total of 18 sessions in 6 weeks.
  Interventions: Device: Sham magnetic stickers; Drug: Chinese herbal medicine

INTERVENTIONS:
Device: Magnetic stickers — 36 patients receive acupoint sticking treatment of Chinese herbal medicine on Dazhui(GV14) and Tiantu(RN22), and magnetic stickers on Feishu(BL13), Pishu(BL20) and Shenshu(BL23) once every other day, retention for 4 hours. Patients receive verum acupoint sticking therapy once every other day with a total of 18 sessions in 6 weeks.
  Other Names: Medical Magnet Points For Aching Pain
  Arms: Acupoint sticking therapy group
Device: Sham magnetic stickers — 36 patients receive acupoint sticking treatment of Chinese herbal medicine on Dazhui(GV14) and Tiantu(RN22), and sham magnetic stickers on Feishu(BL13), Pishu(BL20) and Shenshu(BL23) once every other day, retention for 4 hours. Patients receive verum acupoint sticking therapy once every other day with a total of 18 sessions in 6 weeks.
  Other Names: Blank Points For Aching Pain
  Arms: Sham sticking therapy group
Drug: Chinese herbal medicine — 72 patients receive acupoint sticking treatment of Chinese herbal medicine on Dazhui(GV14) and Tiantu(RN22).
  Other Names: Warm Yang Applicator Party

SUMMARY:
The purpose of this study is to assess whether Acupoint Sticking in Treating Winter Diseases in Summer is effective in the treatment of chronic asthma.

DETAILED DESCRIPTION:
Asthma is a common chronic disease with an estimated 300 million worldwide. Treating Winter Diseases in Summer of traditional Chinese medicine treatment of asthma has a long history. But there are less related clinical trials. The purpose of this study is to assess whether Acupoint Sticking in Treating Winter Diseases in Summer is effective in the treatment of chronic asthma.

After screening period, participants will undergo a physical examination, lung function, blood and induced sputum collection while being randomly assigned to one of the following 2 groups for 6 weeks during summer dog days of treatment:

Group A will receive acupoint sticking treatment of Chinese herbal medicine and magnetic stickers once every two days； Group B will receive acupoint sticking treatment of Chinese herbal medicine and sham magnetic stickers once every two days.

Questionnaires to assess asthma control and quality of life will be completed. A physical examination, blood collection, and induced sputum collection will occur at selected visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with mild-to-moderate remission phase of asthma
* Patients who have given written informed consent

Exclusion Criteria:

* Participation in another clinical trial 1 month prior to study entry
* Participation received acupoint sticking of winter disease cured in summer
* Use of corticosteroids 4 weeks prior to study entry
* Patients who are allergic to therapeutic medicine
* Female patients in lactation period, pregnancy or planning to get pregnant during the trial
* Patients with severe primary diseases such as cancer, cardiovascular system, digestive system, kidney and hematopoietic system diseases
* Patients with mental illness, acrasia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Total score Change from Baseline of Asthma Control Test | Measured during the 6 week treatment period

SECONDARY OUTCOMES:
Cytokine levels of serum and induced sputum | Measured during the 6 week treatment period
Lung function(FEV1, PVC, PEF) | Measured during the 6 week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Zhenhui Lu, doctor, Principal Investigator — Shanghai University of Traditional Chinese Medicine
Locations (1):
- Longhua Hospital Affiliated Shanghai University of TCM, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided